CLINICAL TRIAL: NCT01374516
Title: Efficacy and Safety of a Novel Tetravalent Dengue Vaccine in Healthy Children and Adolescents Aged 9 to 16 Years in Latin America
Brief Title: Study of a Novel Tetravalent Dengue Vaccine in Healthy Children and Adolescents Aged 9 to 16 Years in Latin America
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CYD15; UTN: U1111-1116-4986 (Other: WHO)
Record Dates: First submitted 2011-06-14; First posted 2011-06-16 (Estimated); Results first posted 2019-03-27 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Dengue Fever; Dengue Hemorrhagic Fever; Dengue
Keywords: Dengue Virus; Dengue fever; Dengue Hemorrhagic Fever; CYD dengue vaccine; Flavivirus; Dengue Disease
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CYD Dengue Vaccine Group (Experimental): Participants were to receive 3 doses of CYD dengue vaccine; one each at 0, 6, and 12 months.
  Interventions: Biological: Live, attenuated, dengue serotype 1, 2, 3, 4 virus
- Placebo Group (Placebo Comparator): Participants were to receive a placebo vaccine at 0, 6, and 12 months.
  Interventions: Biological: Placebo: (NaCl) 0.9% solution

INTERVENTIONS:
Biological: Live, attenuated, dengue serotype 1, 2, 3, 4 virus — 0.5 mL, Subcutaneous
  Other Names: CYD Dengue Vaccine
  Arms: CYD Dengue Vaccine Group
Biological: Placebo: (NaCl) 0.9% solution — 0.5 mL, Subcutaneous
  Arms: Placebo Group

SUMMARY:
The aim of the study was to assess the efficacy of Sanofi Pasteur's CYD dengue vaccine in preventing symptomatic virologically-confirmed dengue cases for dengue-endemic areas of Latin America.

Primary Objective:

To assess the efficacy of CYD dengue vaccine after 3 vaccinations at 0, 6, and 12 months in preventing symptomatic virologically-confirmed dengue (VCD) cases, regardless of the severity, due to any of the four serotypes in children and adolescents aged 9 to 16 years at the time of inclusion.

Secondary Objectives:

* To describe the efficacy of CYD dengue vaccine in preventing symptomatic VCD cases after the third dose to the end of the Active Phase, after at least 1 dose, and after 2 doses.
* To describe the occurrence of hospitalized VCD cases and the occurrence of severe (clinically severe or as per World Health Organization (WHO) criteria) VCD cases, throughout the Surveillance Expansion Period (SEP) and throughout the trial (from Day 0 until the end of the study).
* To describe the antibody response to each dengue serotype after Dose 2, after Dose 3, and 1 and 5 years after Dose 3.
* To describe the occurrence of serious adverse events (SAEs), including SAEs of special interest in all participants throughout the trial period.

DETAILED DESCRIPTION:
Participants were randomized to either receive 3 injections of CYD dengue vaccine or a placebo at 0, 6, and 12 months.

A subset of participants from each country (N=2000) was also evaluated for reactogenicity and immunogenicity.

For each participant, the Active Phase of dengue case detection began after the first injection (Dose 1) and continued until 13 months after the third injection (Dose 3). It was assumed that 12 months of surveillance should result in the detection of a sufficient number of VCD cases to allow for an assessment of efficacy.

The Hospital Phase began after the Active Phase. Participants with a febrile illness and requiring hospitalization were screened for dengue until the end of the study.

Participants who consented to participate in the SEP were actively followed for dengue case detection (i.e. at least weekly contact and capturing any acute febrile illness, not just hospitalized febrile cases, as in the Active Phase). The SEP was designed to maximize the detection of symptomatic VCD (hospitalized or not) in order to describe CYD dengue vaccine efficacy and safety in preventing symptomatic dengue in the long-term. Participants who declined participating in the SEP continued surveillance as in the Hospital Phase until trial completion.

Symptomatic VCD cases occurring more than (>) 28 days after dose 3 (during the Active Phase) are defined as:

* Acute febrile illness (i.e. temperature >=38 degree Celsius (°C) on at least 2 consecutive days)
* Virologically confirmed by dengue Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) and/or dengue non-structural (NS)1 enzyme-linked immunosorbent assay (ELISA) Ag test.

Severity was assessed using a definition consistent with the 1997 WHO Classification Dengue Hemorrhagic Fever and by an independent Data Monitoring Committee (IDMC) severity criteria.

ELIGIBILITY:
Inclusion Criteria:

* Aged 9 to 16 years on the day of inclusion and resident of the site zone
* Participant in good health, based on medical history and physical examination
* Assent form or informed consent form has been signed and dated by the participant (based on local regulations), and informed consent form has been signed and dated by the parent(s) or another legally acceptable representative (and by an independent witness if required by local regulations)
* Participant was able to attend all scheduled visits and comply with all trial procedures.

Exclusion Criteria:

* Participant was pregnant, or lactating, or of childbearing potential (to be considered of non-childbearing potential, a female must be pre-menarche for at least 1 year, surgically sterile, or using an effective method of contraception or abstinence from at least 4 weeks prior to the first vaccination until at least 4 weeks after the last vaccination).
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination
* Planned participation in another clinical trial during the present trial period
* Self-reported or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the preceding 6 months; or long-term systemic corticosteroids therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
* Self-reported seropositivity for Human Immunodeficiency Virus (HIV) infection
* Self-reported systemic hypersensitivity to any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the trial or to a vaccine containing any of the same substances
* Chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with trial conduct or completion
* Receipt of blood or blood-derived products in the past 3 months, which might interfere with assessment of the immune response
* Planned receipt of any vaccine in the 4 weeks following any trial vaccination
* Deprived of freedom by administrative or court order, or in an emergency setting, or hospitalized involuntarily
* Current alcohol abuse or drug addiction that may interfere with the participant's ability to comply with trial procedures
* Identified as a site employee of the Investigator or study center, with direct involvement in the proposed study or other studies under the direction of that Investigator or study center, as well as a family member (i.e., immediate, husband, wife and their children, adopted or natural) of the site employees or the Investigator.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20869 (Actual)
Dates: Start 2011-06-08 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2018-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (22):
- Brazil (5):
  - Fortaleza, Ceará
  - Vitória, Espírito Santo
  - Goiânia, Goiás
  - Campo Grande, Mato Grosso do Sul
  - Natal, Rio Grande do Norte
- Colombia (9):
  - Aguazul, Casanare Department
  - Yopal, Casanare Department
  - Girardot City, Cundinamarca
  - Acacías, Meta Department
  - Armenia, Quindío Department
  - Calarcá, Quindío Department
  - La Tebaida, Quindío Department
  - Montenegro, Quindío Department
  - Bucaramanga, Santander Department
- Tegucigalpa, Municipalidad Del Distrito Central, Honduras
- Mexico (5):
  - Temixco, Morelos
  - Municipio de Cd. Mante, Tamaulipas
  - Veracruz Puerto, Veracruz
  - Tizimín, Yucatán
  - Valladolid, Yucatán
- Puerto Rico (2):
  - Guayama
  - San Juan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Result] Villar L, Dayan GH, Arredondo-Garcia JL, Rivera DM, Cunha R, Deseda C, Reynales H, Costa MS, Morales-Ramirez JO, Carrasquilla G, Rey LC, Dietze R, Luz K, Rivas E, Miranda Montoya MC, Cortes Supelano M, Zambrano B, Langevin E, Boaz M, Tornieporth N, Saville M, Noriega F; CYD15 Study Group. Efficacy of a tetravalent dengue vaccine in children in Latin America. N Engl J Med. 2015 Jan 8;372(2):113-23. doi: 10.1056/NEJMoa1411037. Epub 2014 Nov 3. PMID 25365753
- [Result] Hadinegoro SR, Arredondo-Garcia JL, Capeding MR, Deseda C, Chotpitayasunondh T, Dietze R, Muhammad Ismail HI, Reynales H, Limkittikul K, Rivera-Medina DM, Tran HN, Bouckenooghe A, Chansinghakul D, Cortes M, Fanouillere K, Forrat R, Frago C, Gailhardou S, Jackson N, Noriega F, Plennevaux E, Wartel TA, Zambrano B, Saville M; CYD-TDV Dengue Vaccine Working Group. Efficacy and Long-Term Safety of a Dengue Vaccine in Regions of Endemic Disease. N Engl J Med. 2015 Sep 24;373(13):1195-206. doi: 10.1056/NEJMoa1506223. Epub 2015 Jul 27. PMID 26214039
- [Result] Arredondo-Garcia JL, Hadinegoro SR, Reynales H, Chua MN, Rivera Medina DM, Chotpitayasunondh T, Tran NH, Deseda CC, Wirawan DN, Cortes Supelano M, Frago C, Langevin E, Coronel D, Laot T, Perroud AP, Sanchez L, Bonaparte M, Limkittikul K, Chansinghakul D, Gailhardou S, Noriega F, Wartel TA, Bouckenooghe A, Zambrano B; CYD-TDV Dengue Vaccine Study Group. Four-year safety follow-up of the tetravalent dengue vaccine efficacy randomized controlled trials in Asia and Latin America. Clin Microbiol Infect. 2018 Jul;24(7):755-763. doi: 10.1016/j.cmi.2018.01.018. Epub 2018 Feb 8. PMID 29408333
- [Result] L'Azou M, Moureau A, Sarti E, Nealon J, Zambrano B, Wartel TA, Villar L, Capeding MR, Ochiai RL; CYD14 Primary Study Group; CYD15 Primary Study Group. Symptomatic Dengue in Children in 10 Asian and Latin American Countries. N Engl J Med. 2016 Mar 24;374(12):1155-66. doi: 10.1056/NEJMoa1503877. PMID 27007959
- [Result] Sridhar S, Luedtke A, Langevin E, Zhu M, Bonaparte M, Machabert T, Savarino S, Zambrano B, Moureau A, Khromava A, Moodie Z, Westling T, Mascarenas C, Frago C, Cortes M, Chansinghakul D, Noriega F, Bouckenooghe A, Chen J, Ng SP, Gilbert PB, Gurunathan S, DiazGranados CA. Effect of Dengue Serostatus on Dengue Vaccine Safety and Efficacy. N Engl J Med. 2018 Jul 26;379(4):327-340. doi: 10.1056/NEJMoa1800820. Epub 2018 Jun 13. PMID 29897841
- [Derived] Savarino SJ, Bonaparte M, Wang H, Dayan GH, Forrat R, Zhu M, Hodge S, Ataman-Onal Y, DiazGranados CA. Accuracy and efficacy of pre-dengue vaccination screening for previous dengue infection with a new dengue rapid diagnostic test: a retrospective analysis of phase 3 efficacy trials. Lancet Microbe. 2022 Jun;3(6):e427-e434. doi: 10.1016/S2666-5247(22)00033-7. Epub 2022 May 4. PMID 35659904
- [Derived] Laydon DJ, Dorigatti I, Hinsley WR, Nedjati-Gilani G, Coudeville L, Ferguson NM. Efficacy profile of the CYD-TDV dengue vaccine revealed by Bayesian survival analysis of individual-level phase III data. Elife. 2021 Jul 2;10:e65131. doi: 10.7554/eLife.65131. PMID 34219653
- [Derived] Henein S, Adams C, Bonaparte M, Moser JM, Munteanu A, Baric R, de Silva AM. Dengue vaccine breakthrough infections reveal properties of neutralizing antibodies linked to protection. J Clin Invest. 2021 Jul 1;131(13):e147066. doi: 10.1172/JCI147066. PMID 34003796
- [Derived] Forrat R, Dayan GH, DiazGranados CA, Bonaparte M, Laot T, Capeding MR, Sanchez L, Coronel DL, Reynales H, Chansinghakul D, Hadinegoro SRS, Perroud AP, Frago C, Zambrano B, Machabert T, Wu Y, Luedtke A, Price B, Vigne C, Haney O, Savarino SJ, Bouckenooghe A, Noriega F. Analysis of Hospitalized and Severe Dengue Cases Over the 6 years of Follow-up of the Tetravalent Dengue Vaccine (CYD-TDV) Efficacy Trials in Asia and Latin America. Clin Infect Dis. 2021 Sep 15;73(6):1003-1012. doi: 10.1093/cid/ciab288. PMID 33822015
- [Derived] DiazGranados CA, Bonaparte M, Wang H, Zhu M, Lustig Y, Schwartz E, Forrat R, Dayan GH, Hodge S, Ataman-Onal Y, Savarino SJ. Accuracy and efficacy of pre-dengue vaccination screening for previous dengue infection with five commercially available immunoassays: a retrospective analysis of phase 3 efficacy trials. Lancet Infect Dis. 2021 Apr;21(4):529-536. doi: 10.1016/S1473-3099(20)30695-2. Epub 2020 Nov 16. PMID 33212068
- [Derived] Reynales H, Carrasquilla G, Zambrano B, Cortes S M, Machabert T, Jing J, Pallardy S, Haney O, Faccini M, Quintero J, Noriega F. Secondary Analysis of the Efficacy and Safety Trial Data of the Tetravalent Dengue Vaccine in Children and Adolescents in Colombia. Pediatr Infect Dis J. 2020 Apr;39(4):e30-e36. doi: 10.1097/INF.0000000000002580. PMID 32040014
- [Derived] Plennevaux E, Moureau A, Arredondo-Garcia JL, Villar L, Pitisuttithum P, Tran NH, Bonaparte M, Chansinghakul D, Coronel DL, L'Azou M, Ochiai RL, Toh ML, Noriega F, Bouckenooghe A. Impact of Dengue Vaccination on Serological Diagnosis: Insights From Phase III Dengue Vaccine Efficacy Trials. Clin Infect Dis. 2018 Apr 3;66(8):1164-1172. doi: 10.1093/cid/cix966. PMID 29300876
- [Derived] Rabaa MA, Girerd-Chambaz Y, Duong Thi Hue K, Vu Tuan T, Wills B, Bonaparte M, van der Vliet D, Langevin E, Cortes M, Zambrano B, Dunod C, Wartel-Tram A, Jackson N, Simmons CP. Genetic epidemiology of dengue viruses in phase III trials of the CYD tetravalent dengue vaccine and implications for efficacy. Elife. 2017 Sep 5;6:e24196. doi: 10.7554/eLife.24196. PMID 28871961
- [Derived] Harenberg A, de Montfort A, Jantet-Blaudez F, Bonaparte M, Boudet F, Saville M, Jackson N, Guy B. Cytokine Profile of Children Hospitalized with Virologically-Confirmed Dengue during Two Phase III Vaccine Efficacy Trials. PLoS Negl Trop Dis. 2016 Jul 26;10(7):e0004830. doi: 10.1371/journal.pntd.0004830. eCollection 2016 Jul. PMID 27459266
- [Derived] Olivera-Botello G, Coudeville L, Fanouillere K, Guy B, Chambonneau L, Noriega F, Jackson N; CYD-TDV Vaccine Trial Group. Tetravalent Dengue Vaccine Reduces Symptomatic and Asymptomatic Dengue Virus Infections in Healthy Children and Adolescents Aged 2-16 Years in Asia and Latin America. J Infect Dis. 2016 Oct 1;214(7):994-1000. doi: 10.1093/infdis/jiw297. Epub 2016 Jul 14. PMID 27418050
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 08 June 2011 to 16 March 2012 at 5 clinical centers in Brazil, 9 in Colombia, 1 in Honduras, 5 in Mexico, and 2 in Puerto Rico.
Pre-assignment Details: A total of 20869 participants were enrolled and randomized in the study.
Groups:
- CYD Dengue Vaccine Group: Participants received 3 doses of CYD dengue vaccine; one each at 0, 6, and 12 months and were followed up to 60 months after last vaccination (or a total duration of up to 72 months).
- Placebo Group: Participants received 3 doses of placebo matched to vaccine; one each at 0, 6, and 12 months and were followed up to 60 months after last vaccination (or a total duration of up to 72 months).
Period: Vaccination Phase (Up to 25 Months)
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Started | 13920 | 6949
Completed | 13281 | 6640
Not Completed | 639 | 309
Not completed — Protocol Violation | 43 | 14
Not completed — Adverse Event | 3 | 0
Not completed — Withdrawal by Subject | 480 | 240
Not completed — Lost to Follow-up | 106 | 46
Not completed — Serious adverse event | 7 | 9
Period: Surveillance Expansion Period
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Started | 13281 | 6640
Completed | 10932 | 5387
Not Completed | 2349 | 1253
Not completed — Protocol Violation | 386 | 217
Not completed — Withdrawal by Subject | 1870 | 986
Not completed — Lost to Follow-up | 73 | 45
Not completed — Serious adverse event | 20 | 5

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine Group | Placebo Group | Total
Number analyzed (Participants) | 13920 | 6949 | 20869
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13920 | 6949 | 20869
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years]
  Age Continuous | 12.5 (2.14) | 12.5 (2.13) | 12.5 (2.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7048 | 3532 | 10580
  Male | 6872 | 3417 | 10289
Region of Enrollment [Number; unit: Participants]
  Colombia | 6497 | 3246 | 9743
  Brazil | 2370 | 1178 | 3548
  Mexico | 2312 | 1152 | 3464
  Honduras | 1866 | 933 | 2799
  Puerto Rico | 875 | 440 | 1315

OUTCOME MEASURES:

1. Primary Outcome: Number of Symptomatic Virologically Confirmed Dengue (VCD) Cases Due to Any Serotype During the Active Phase Post-dose 3 Following Injection With Either CYD Dengue Vaccine or a Placebo
Description: Symptomatic VCD cases were defined as occurrence of acute febrile illness (temperature >=38°C on at least 2 consecutive days) and confirmation of dengue virus infection by dengue reverse transcriptase polymerase chain reaction (RT-PCR) and/or dengue non-structural (NS) protein 1 antigen enzyme-linked immunosorbent assay (ELISA). Vaccine efficacy was defined as 1 minus the ratio of density incidence due to any serotype after at least 1 dose in the CYD Dengue Vaccine Group over the density incidence of the Placebo Group.
Time Frame: 28 days and up to 13 months post-injection 3
Population: Number of symptomatic VCD cases were assessed in the Per-Protocol Analysis Set for Efficacy, defined as participants who had no protocol deviations.
Measure: Number; unit: Cases
Groups:
- CYD Dengue Vaccine Group: Participants received 3 doses of CYD dengue vaccine; one each at 0, 6, and 12 months.
- Placebo Group: Participants received 3 doses of placebo matched to vaccine; one each at 0, 6, and 12 months.
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 12574 | 6261
Cases | 176 | 221
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Placebo Group; The statistical methodology was based on the use of the two-sided 95% confidence interval (CI) of the vaccine efficacy (expressed in %). The CI was calculated using the exact method conditional on the total number of cases in both groups (exact method by Breslow & Day). The vaccine efficacy of the CYD dengue vaccine was considered significant if the lower bound of its 95% CI was greater than 25%; Test type: Superiority or Other; Vaccine Efficacy = 60.8, 95% CI 2-sided [52.0 to 68.0]

2. Secondary Outcome: Number of Symptomatic VCD Cases Due to Any Serotype During the Active Phase Following Injection With Either CYD Dengue Vaccine or a Placebo
Description: Symptomatic VCD cases were defined as occurrence of acute febrile illness (temperature >=38°C on at least 2 consecutive days) and confirmation of dengue virus infection by dengue RT-PCR and/or dengue NS 1 ELISA. Vaccine efficacy was defined as 1 minus the ratio of density incidence due to any serotype after at least 1 dose in the CYD Dengue Vaccine Group over the density incidence of the Placebo Group.
Time Frame: Day 0 up to 13 months post-injection 3
Population: Number of symptomatic VCD cases were assessed in the Full Analysis Set for Efficacy, which included all participants who received at least 1 injection.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 13914 | 6940
Cases | 277 | 385
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Placebo Group; The statistical methodology was based on the use of the two-sided 95% CI of the vaccine efficacy (expressed in %) calculated using the exact method conditional on the total number of cases in both groups; Test type: Superiority or Other; Vaccine Efficacy = 64.7, 95% CI 2-sided [58.7 to 69.8]

3. Secondary Outcome: Number of Symptomatic VCD Cases Due to Any Serotype Occurring 28 Days Post-dose 1 Following Injection With Either CYD Dengue Vaccine or a Placebo
Description: Symptomatic VCD cases were defined as occurrence of acute febrile illness (temperature >= 38°C on at least 2 consecutive days) and confirmation of dengue virus infection by dengue RT-PCR and/or dengue NS 1 ELISA. Vaccine efficacy was defined as 1 minus the ratio of density incidence due to any serotype after at least 1 dose in the CYD Dengue Vaccine Group over the density incidence of the Placebo Group.
Time Frame: 28 days post-injection 1 and up to 13 months post-injection 3
Population: Number of symptomatic VCD cases were assessed in the Full Analysis Set for Efficacy, which included participants who received at least 1 dose of study vaccine.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 13914 | 6940
Cases | 273 | 380
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Placebo Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Vaccine Efficacy = 64.7, 95% CI 2-sided [58.7 to 69.9]

4. Secondary Outcome: Number of Symptomatic VCD Cases Due to Any Serotype Post-dose 2 Following Injection With Either CYD Dengue Vaccine or a Placebo
Description: as for outcome 3
Time Frame: 28 days post-injection 2 and up to 13 months post-injection 3
Population: Number of symptomatic VCD cases were assessed in the Other Efficacy Analysis Set, which included participants who received at least 2 doses of study vaccine.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 13506 | 6765
Cases | 236 | 306
Statistical Analysis 1: Comparison: CYD Dengue Vaccine Group vs Placebo Group; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; Vaccine Efficacy = 61.9, 95% CI 2-sided [54.7 to 68.0]

5. Secondary Outcome: Number of Symptomatic VCD Cases Meeting World Health Organization (WHO) Criteria Throughout the Trial Due to Any Serotype Following Injection With Either CYD Dengue Vaccine or a Placebo
Description: Dengue hemorrhagic fever (DHF) cases were defined as number of participants with at least one symptomatic VCD episode meeting the 1997 WHO criteria. (a) Fever: acute onset, high (>= 38°C) and continuous, lasting 2 to 7 days and (b) any of the pre-listed hemorrhagic manifestations and laboratory findings of thrombocytopenia (platelet <=100 x 109/L) and plasma leakage as shown by hemoconcentration (hematocrit increased by 20% or more) or pleural effusion (seen on CXR) and/or ascites and/ or hypoalbuminemia. The first two clinical criteria plus thrombocytopenia and signs of plasma leakage are enough to establish a clinical diagnosis of DHF. DHF was graded as follows: Grade I: Fever accompanied by non-specific constitutional symptoms; the only hemorrhagic manifestation is a positive tourniquet test; Grade II: Spontaneous bleeding in addition to the manifestations of Grade I participants, usually in the form of skin and/or other hemorrhage.
Time Frame: Day 0 to the end of study (up to 72 months)
Population: Number of WHO dengue hemorrhagic fever cases were assessed in the Safety Analysis Set, which included all participants who received at least one dose of study vaccine. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 12809 | 6380
Cases
  Due to Any of the 4 Serotypes: Any Grade | 7 | 15
  Due to Any of the 4 Serotypes: Grade I | 0 | 2
  Due to Any of the 4 Serotypes: Grade II | 7 | 13
  Due to Any of the 4 Serotypes: Grade III | 0 | 0
  Due to Any of the 4 Serotypes: Grade IV | 0 | 0

6. Secondary Outcome: Number of Symptomatic VCD Cases Meeting WHO Criteria During the Surveillance Expansion Period Due to Any Serotype Following Injection With Either CYD Dengue Vaccine or a Placebo
Description: The 1997 WHO criteria are: a) Fever: acute onset, high (>= 38°C) and continuous, for 2 to 7 days and (b) any of the following: thrombocytopenia (platelet <=100 x 109/L) and plasma leakage as shown by hematocrit increased by 20% or more or pleural effusion and/or ascites and/or hypoalbuminemia. The first two clinical criteria plus thrombocytopenia and signs of plasma leakage are enough to establish diagnosis of DHF. DHF was graded as follows: Grade I: Fever accompanied by non-specific constitutional symptoms; the only hemorrhagic manifestation is a positive tourniquet test; Grade II: Spontaneous bleeding in addition to the manifestations of Grade I participant, usually in the form of skin and/or other hemorrhages; Grade III: Circulatory failure manifested by rapid and weak pulse, narrowing of pulse pressure (20 mmHg or less) or hypotension, with the presence of cold clammy skin and restlessness; and Grade IV: Profound shock with undetectable blood pressure and pulse.
Time Frame: From consent to participate in the Surveillance Expansion Period to the end of study (up to 72 months)
Population: Number of WHO dengue hemorrhagic fever cases were assessed in the Full Analysis Set for Surveillance Expansion Period, which included all participants who received at least 1 injection and accepted to be included in the Surveillance Expansion Period.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 11063 | 5430
Cases
  Due to Any of the 4 Serotypes: Any Grade | 2 | 0
  Due to Any of the 4 Serotypes: Grade I | 0 | 0
  Due to Any of the 4 Serotypes: Grade II | 2 | 0
  Due to Any of the 4 Serotypes: Grade III | 0 | 0
  Due to Any of the 4 Serotypes: Grade IV | 0 | 0

7. Secondary Outcome: Number of Hospitalized VCD Cases Throughout the Trial Due to Any Serotype Following Injection With Either CYD Dengue Vaccine or a Placebo
Description: Hospitalized VCD cases were defined as VCD confirmed by dengue RT-PCR and/or dengue NS 1 ELISA in participants with acute febrile illness (temperature >=38°C on at least 2 consecutive days) requiring hospitalization.
Time Frame: Day 0 up to the end of study (up to 72 months)
Population: Number of hospitalized dengue hemorrhagic fever cases were assessed in the Safety Analysis Set. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 12809 | 6380
Cases | 46 | 71

8. Secondary Outcome: Number of Hospitalized VCD Cases During the Surveillance Expansion Period Due to Any Serotype Following Injection With Either CYD Dengue Vaccine or a Placebo
Description: as for outcome 7
Time Frame: From consent to participate in the Surveillance Expansion Period to end of the study (up to 72 months)
Population: Analysis was performed in the Safety Analysis Set.
Measure: Number; unit: Cases
Groups:
- Control Group: Participants received 3 doses of placebo matched to vaccine; one each at 0, 6, and 12 months and were followed up to 60 months after last vaccination (or a total duration of up to 72 months).
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 13915 | 6939
Cases | 5 | 2

9. Secondary Outcome: Number of Clinically Severe VCD Cases Throughout the Trial Due to Any Serotype Following Injection With Either CYD Dengue Vaccine or a Placebo
Description: The severity of VCD cases was assessed by an Independent Data monitoring Committee (IDMC) based on a medical review of cases and any of the following criteria:1) Platelet count <=100000 /μl and bleeding (tourniquet, petechiae or any bleeding) plus plasma leakage 2) Shock (pulse pressure <= 20 mmHg in a child, or hypotension [<= 90 mmHg] with tachycardia, weak pulse and poor perfusion) 3) Bleeding requiring blood transfusion 4) Encephalopathy i.e. unconsciousness or poor conscious state or fitting not attributable to simple febrile convulsion or focal neurological signs. Poor conscious state or unconsciousness must be supported by Glasgow Coma Scale (GCS) score 5) Liver impairment (AST >1000 IU/L or prothrombin time [PT] International normalized ratio [INR] >1.5) excluding other causes of viral hepatitis 6) Impaired kidney function (serum creatinine >= 1.5 mg/dL) 7) Myocarditis, pericarditis or clinical heart failure supported by CXR, echocardiography, ECG or cardiac enzymes.
Time Frame: Day 0 to the end of study (up to 72 months)
Population: Number of clinically severe VCD cases were assessed in the Safety Analysis Set. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 12809 | 6380
Cases | 9 | 16

10. Secondary Outcome: Number of Clinically Severe VCD Cases During the Surveillance Expansion Period Due to Any Serotype Following Injection With Either CYD Dengue Vaccine or a Placebo
Description: The severity of VCD cases was assessed by an IDMC based on a medical review of cases and any of the following criteria:-1) Platelet count <=100000 /μl and bleeding (tourniquet, petechiae or any bleeding) plus plasma leakage 2) Shock (pulse pressure <= 20 mmHg in a child, or hypotension [<= 90 mmHg] with tachycardia, weak pulse and poor perfusion) 3) Bleeding requiring blood transfusion 4) Encephalopathy i.e. Unconsciousness or poor conscious state or fitting not attributable to simple febrile convulsion or focal neurological signs. Poor conscious state or unconsciousness must be supported by GCS score 5) Liver impairment (AST >1000 IU/L or PT INR >1.5) excluding other causes of viral hepatitis 6) Impaired kidney function (serum creatinine >= 1.5 mg/dL) 7) Myocarditis, pericarditis or clinical heart failure supported by CXR, echocardiography, ECG or cardiac enzymes.
Time Frame: From consent to participate in the Surveillance Expansion Period to the end of study (up to 72 months)
Population: Number of clinically severe VCD cases were assessed in the Full Analysis Set for Surveillance Expansion Period. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Number; unit: Cases
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 11061 | 5431
Cases | 42 | 34

11. Secondary Outcome: Percentage of Participants With Antibody Titers >=10 1/Dil Against Each Dengue Virus Serotype Before and Following Injection (Inj.) With CYD Dengue Vaccine or Placebo
Description: Dengue neutralizing antibody levels against each of the 4 dengue virus serotypes (parental strains) were measured by the plaque reduction neutralization test in a pre-defined subset of participants.
Time Frame: Pre-injection 1, 28 days post Injections 2 and 3, 13 months (Visit [V] 07) and 60 months (Visit [V] 12) post-injection 3
Population: Antibody titers against each dengue virus serotype strain were assessed in Full Analysis Set for Immunogenicity(FASI),which included a subset of participants who received at least one dose of vaccine and had a blood sample drawn and result available after the dose.Here, 'number analyzed'=participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Groups:
- CYD Dengue Vaccine Group: Subset of participants who received at least one dose of CYD Dengue vaccine.
- Placebo Group: Subset of participants who received at least one dose of placebo vaccine.
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 1301 | 643
Percentage of participants
  Dengue virus Serotype 1: Pre-Inj.1: number analyzed (Participants) | 1297 | 641
  Dengue virus Serotype 1: Pre-Inj.1 | 72.8 | 70.5
  Dengue virus Serotype 1: Post-Inj. 2: number analyzed (Participants) | 1296 | 638
  Dengue virus Serotype 1: Post-Inj. 2 | 92.7 | 71.8
  Dengue virus Serotype 1: Post-Inj. 3: number analyzed (Participants) | 1291 | 640
  Dengue virus Serotype 1: Post-Inj. 3 | 94.9 | 74.2
  Dengue virus Serotype 1; 1 year Post-Inj. 3 (V 07): number analyzed (Participants) | 1261 | 629
  Dengue virus Serotype 1; 1 year Post-Inj. 3 (V 07) | 85.6 | 73.6
  Dengue virus Serotype 1; 5 year Post-Inj. 3 (V 12): number analyzed (Participants) | 1038 | 508
  Dengue virus Serotype 1; 5 year Post-Inj. 3 (V 12) | 90.0 | 81.1
  Dengue virus Serotype 2; Pre-Inj. 1: number analyzed (Participants) | 1299 | 640
  Dengue virus Serotype 2; Pre-Inj. 1 | 76.1 | 73.8
  Dengue virus Serotype 2; Post-Inj. 2: number analyzed (Participants) | 1297 | 639
  Dengue virus Serotype 2; Post-Inj. 2 | 97.5 | 75.1
  Dengue virus Serotype 2; Post-Inj. 3: number analyzed (Participants) | 1291 | 640
  Dengue virus Serotype 2; Post-Inj. 3 | 98.5 | 77.2
  Dengue virus Serotype 2; 1 year Post-Inj. 3 (V 07): number analyzed (Participants) | 1264 | 629
  Dengue virus Serotype 2; 1 year Post-Inj. 3 (V 07) | 94.1 | 78.9
  Dengue virus Serotype 2; 5 year Post-Inj. 3 (V 12): number analyzed (Participants) | 1038 | 508
  Dengue virus Serotype 2; 5 year Post-Inj. 3 (V 12) | 93.5 | 83.1
  Dengue virus Serotype 3; Pre-Inj. 1: number analyzed (Participants) | 1300 | 639
  Dengue virus Serotype 3; Pre-Inj. 1 | 76.5 | 73.6
  Dengue virus Serotype 3; Post-Inj. 2: number analyzed (Participants) | 1297 | 639
  Dengue virus Serotype 3; Post-Inj. 2 | 98.5 | 75.7
  Dengue virus Serotype 3; Post-Inj. 3: number analyzed (Participants) | 1291 | 640
  Dengue virus Serotype 3; Post-Inj. 3 | 98.4 | 78.0
  Dengue virus Serotype 3; 1 year Post-Inj. 3 (V 07): number analyzed (Participants) | 1265 | 629
  Dengue virus Serotype 3; 1 year Post-Inj. 3 (V 07) | 92.7 | 76.2
  Dengue virus Serotype 3; 5 year Post-Inj. 3 (V 12): number analyzed (Participants) | 1038 | 508
  Dengue virus Serotype 3; 5 year Post-Inj. 3 (V 12) | 95.4 | 82.7
  Dengue virus Serotype 4; Pre-Inj. 1: number analyzed (Participants) | 1297 | 640
  Dengue virus Serotype 4; Pre-Inj. 1 | 68.2 | 65.0
  Dengue virus Serotype 4; Post-Inj. 2: number analyzed (Participants) | 1295 | 637
  Dengue virus Serotype 4; Post-Inj. 2 | 96.9 | 67.0
  Dengue virus Serotype 4; Post-Inj. 3: number analyzed (Participants) | 1291 | 640
  Dengue virus Serotype 4; Post-Inj. 3 | 98.1 | 68.9
  Dengue virus Serotype 4; 1 year Post-Inj. 3 (V 07): number analyzed (Participants) | 1265 | 625
  Dengue virus Serotype 4; 1 year Post-Inj. 3 (V 07) | 94.9 | 69.0
  Dengue virus Serotype 4; 5 year Post-Inj. 3 (V 12): number analyzed (Participants) | 1038 | 508
  Dengue virus Serotype 4; 5 year Post-Inj. 3 (V 12) | 96.3 | 78.9

12. Secondary Outcome: Geometric Mean Titers of Antibodies Against Each Dengue Virus Serotype Before and Following Injection With Either CYD Dengue Tetravalent Vaccine or a Placebo
Description: Geometric mean titers for each of the 4 dengue virus serotypes (parental strains) were assessed using the plaque reduction neutralization test in a pre-defined subset of participants.
Time Frame: Pre-injection 1, 28 days post Injections 2 and 3, 13 months (V 07) and 60 months (V 12) post-injection 3
Population: Antibody titers against each dengue virus serotype strain were assessed in FASI, which included a subset of participants who received at least one dose of vaccine and had a blood sample drawn and result available after the dose. Here,'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dilution)
Groups:
- Placebo Group: Subset of participants who received at least one dose of the placebo vaccine.
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 1301 | 643
Titers (1/dilution)
  Dengue virus Serotype 1; Pre-Inj. 1: number analyzed (Participants) | 1297 | 641
  Dengue virus Serotype 1; Pre-Inj. 1 | 128 [112 to 145] | 119 [98.7 to 142]
  Dengue virus Serotype 1; Post Inj. 2: number analyzed (Participants) | 1296 | 638
  Dengue virus Serotype 1; Post Inj. 2 | 458 [406 to 517] | 128 [106 to 154]
  Dengue virus Serotype 1; Post Inj. 3: number analyzed (Participants) | 1291 | 640
  Dengue virus Serotype 1; Post Inj. 3 | 395 [353 to 441] | 121 [101 to 145]
  Dengue virus Serotype 1; Year 1 Post Inj. 3 (V 07): number analyzed (Participants) | 1261 | 629
  Dengue virus Serotype 1; Year 1 Post Inj. 3 (V 07) | 266 [234 to 302] | 146 [121 to 176]
  Dengue virus Serotype 1; Year 5 Post Inj. 3 (V 12): number analyzed (Participants) | 1038 | 508
  Dengue virus Serotype 1; Year 5 Post Inj. 3 (V 12) | 284 [252 to 321] | 210 [172 to 255]
  Dengue virus Serotype 2; Pre-Inj. 1: number analyzed (Participants) | 1299 | 640
  Dengue virus Serotype 2; Pre-Inj. 1 | 138 [123 to 156] | 115 [97.2 to 136]
  Dengue virus Serotype 2; Post Inj. 2: number analyzed (Participants) | 1297 | 639
  Dengue virus Serotype 2; Post Inj. 2 | 622 [566 to 684] | 124 [104 to 148]
  Dengue virus Serotype 2; Post Inj. 3: number analyzed (Participants) | 1291 | 640
  Dengue virus Serotype 2; Post Inj. 3 | 574 [528 to 624] | 129 [109 to 152]
  Dengue virus Serotype 2; Year 1 Post-Inj. 3 (V 07): number analyzed (Participants) | 1264 | 629
  Dengue virus Serotype 2; Year 1 Post-Inj. 3 (V 07) | 371 [336 to 409] | 145 [122 to 173]
  Dengue virus Serotype 2; Year 5 Post-Inj. 3 (V 12): number analyzed (Participants) | 1038 | 508
  Dengue virus Serotype 2; Year 5 Post-Inj. 3 (V 12) | 297 [269 to 328] | 201 [168 to 242]
  Dengue virus Serotype 3; Pre-Inj. 1: number analyzed (Participants) | 1300 | 639
  Dengue virus Serotype 3; Pre-Inj. 1 | 121 [108 to 136] | 114 [95.9 to 136]
  Dengue virus Serotype 3; Post Inj. 2: number analyzed (Participants) | 1297 | 639
  Dengue virus Serotype 3; Post Inj. 2 | 556 [506 to 610] | 117 [98.3 to 139]
  Dengue virus Serotype 3; Post Inj. 3: number analyzed (Participants) | 1291 | 640
  Dengue virus Serotype 3; Post Inj. 3 | 508 [465 to 555] | 124 [105 to 147]
  Dengue virus Serotype 3; Year 1 Post Inj. 3 (V 07): number analyzed (Participants) | 1265 | 629
  Dengue virus Serotype 3; Year 1 Post Inj. 3 (V 07) | 292 [263 to 325] | 137 [114 to 165]
  Dengue virus Serotype 3; Year 5 Post Inj. 3 (V 12): number analyzed (Participants) | 1038 | 508
  Dengue virus Serotype 3; Year 5 Post Inj. 3 (V 12) | 346 [313 to 383] | 224 [185 to 271]
  Dengue virus Serotype 4; Pre Inj. 1: number analyzed (Participants) | 1297 | 640
  Dengue virus Serotype 4; Pre Inj. 1 | 43.6 [39.6 to 48.0] | 39.0 [33.9 to 44.7]
  Dengue virus Serotype 4; Post Inj. 2: number analyzed (Participants) | 1295 | 637
  Dengue virus Serotype 4; Post Inj. 2 | 261 [242 to 281] | 40.9 [35.5 to 47.0]
  Dengue virus Serotype 4; Post Inj. 3: number analyzed (Participants) | 1291 | 640
  Dengue virus Serotype 4; Post Inj. 3 | 241 [226 to 258] | 44.3 [38.6 to 50.8]
  Dengue virus Serotype 4; Year 1 Post Inj. 3 (V 07): number analyzed (Participants) | 1265 | 625
  Dengue virus Serotype 4; Year 1 Post Inj. 3 (V 07) | 174 [161 to 188] | 51.5 [44.3 to 59.8]
  Dengue virus Serotype 4; Year 5 Post Inj. 3 (V 12): number analyzed (Participants) | 1038 | 508
  Dengue virus Serotype 4; Year 5 Post Inj. 3 (V 12) | 144 [134 to 156] | 73.6 [63.4 to 85.5]

13. Secondary Outcome: Number of Participants With Solicited Injection Site Reactions Following Any and Each Injection With Either CYD Dengue Vaccine or a Placebo
Description: Solicited injection site reactions: Pain, Erythema, and Swelling. Grade 3 reactions (9-11 years): Pain: incapacitating, unable to perform usual activities; Erythema and Swelling, >= 50 mm. Grade 3 Solicited injection site reactions (12-16 years): Pain: significant, prevents daily activity; Erythema and Swelling, >100 mm.
Time Frame: Within 7 days after each and any injection
Population: Solicited injection site reactions were assessed in a subset of the Safety Analysis Set, which included all participants who received at least one dose of study vaccine and who were evaluated for reactogenicity. Here, 'number analyzed' = participants with available data for specified category.
Measure: Number; unit: Participants
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
Number analyzed (Participants) | 1333 | 664
Participants
  Injection-site Pain (Post any injection): number analyzed (Participants) | 1328 | 658
  Injection-site Pain (Post any injection) | 650 | 270
  Injection-site Erythema (Post-any injection): number analyzed (Participants) | 1328 | 658
  Injection-site Erythema (Post-any injection) | 83 | 44
  Injection-site Swelling (Post-any injection): number analyzed (Participants) | 1328 | 658
  Injection-site Swelling (Post-any injection) | 77 | 27
  Injection-site Pain (Post-injection 1): number analyzed (Participants) | 1326 | 657
  Injection-site Pain (Post-injection 1) | 430 | 173
  Grade 3 Injection-site Pain (Post-injection 1): number analyzed (Participants) | 1326 | 657
  Grade 3 Injection-site Pain (Post-injection 1) | 11 | 6
  Injection-site Erythema (Post-injection 1): number analyzed (Participants) | 1326 | 656
  Injection-site Erythema (Post-injection 1) | 55 | 31
  Grade 3 Injection-site Erythema (Post-injection 1): number analyzed (Participants) | 1326 | 656
  Grade 3 Injection-site Erythema (Post-injection 1) | 0 | 1
  Injection-site Swelling (Post-injection 1): number analyzed (Participants) | 1326 | 656
  Injection-site Swelling (Post-injection 1) | 47 | 18
  Grade 3 Injection-site Swelling (Post-injection 1): number analyzed (Participants) | 1326 | 656
  Grade 3 Injection-site Swelling (Post-injection 1) | 0 | 1
  Injection-site Pain (Post-injection 2): number analyzed (Participants) | 1297 | 639
  Injection-site Pain (Post-injection 2) | 332 | 105
  Grade 3 Injection-site Pain (Post-injection 2): number analyzed (Participants) | 1297 | 639
  Grade 3 Injection-site Pain (Post-injection 2) | 7 | 0
  Injection-site Erythema (Post-injection 2): number analyzed (Participants) | 1296 | 639
  Injection-site Erythema (Post-injection 2) | 25 | 11
  Grade 3 Injection-site Erythema (Post-injection 2): number analyzed (Participants) | 1296 | 639
  Grade 3 Injection-site Erythema (Post-injection 2) | 1 | 0
  Injection-site Swelling (Post-injection 2): number analyzed (Participants) | 1296 | 639
  Injection-site Swelling (Post-injection 2) | 25 | 6
  Grade 3 Injection-site Swelling (Post-injection 2): number analyzed (Participants) | 1296 | 639
  Grade 3 Injection-site Swelling (Post-injection 2) | 0 | 0
  Injection-site Pain (Post-injection 3): number analyzed (Participants) | 1279 | 630
  Injection-site Pain (Post-injection 3) | 288 | 104
  Grade 3 Injection-site Pain (Post-injection 3): number analyzed (Participants) | 1279 | 630
  Grade 3 Injection-site Pain (Post-injection 3) | 11 | 2
  Injection-site Erythema (Post-injection 3): number analyzed (Participants) | 1278 | 631
  Injection-site Erythema (Post-injection 3) | 19 | 10
  Grade 3 Injection-site Erythema (Post-injection 3): number analyzed (Participants) | 1278 | 631
  Grade 3 Injection-site Erythema (Post-injection 3) | 0 | 0
  Injection-site Swelling (Post-injection 3): number analyzed (Participants) | 1279 | 631
  Injection-site Swelling (Post-injection 3) | 20 | 8
  Grade 3 Injection-site Swelling (Post-injection 3): number analyzed (Participants) | 1279 | 631
  Grade 3 Injection-site Swelling (Post-injection 3) | 0 | 0

14. Secondary Outcome: Number of Participants With Solicited Systemic Reactions Following Any and Each Injection With Either CYD Dengue Vaccine or a Placebo
Description: Solicited systemic reactions: Fever (Temperature), Headache, Malaise, Myalgia, and Asthenia. Grade 3 reactions: Fever: >= 39°C; Headache, Malaise, Myalgia, and Asthenia: significant, prevents daily activity.
Time Frame: Within 14 days after each and any injection
Population: Solicited systemic reactions were assessed in a subset of the Safety Analysis Set, which included all participants who received at least one dose of study vaccine and who were evaluated for reactogenicity. Here, 'number analyzed' = participants with available data for specified category.
Measure: Number; unit: Participants
Groups:
- Control Group: Participants received 3 doses of placebo matched to vaccine; one each at 0, 6, and 12 months.
Arm/Group | CYD Dengue Vaccine Group | Control Group
Number analyzed (Participants) | 1333 | 664
Participants
  Fever (Post any injection): number analyzed (Participants) | 1318 | 654
  Fever (Post any injection) | 220 | 123
  Headache (Post any injection): number analyzed (Participants) | 1328 | 659
  Headache (Post any injection) | 727 | 379
  Malaise (Post any injection): number analyzed (Participants) | 1328 | 659
  Malaise (Post any injection) | 536 | 261
  Myalgia (Post any injection): number analyzed (Participants) | 1328 | 659
  Myalgia (Post any injection) | 576 | 267
  Asthenia (Post any injection): number analyzed (Participants) | 1328 | 659
  Asthenia (Post any injection) | 496 | 251
  Fever (Post-injection 1): number analyzed (Participants) | 1264 | 635
  Fever (Post-injection 1) | 86 | 42
  Grade 3 Fever (Post-injection 1): number analyzed (Participants) | 1264 | 635
  Grade 3 Fever (Post-injection 1) | 21 | 7
  Headache (Post-injection 1): number analyzed (Participants) | 1324 | 657
  Headache (Post-injection 1) | 528 | 273
  Grade 3 Headache (Post-injection 1): number analyzed (Participants) | 1324 | 657
  Grade 3 Headache (Post-injection 1) | 67 | 27
  Malaise (Post-injection 1): number analyzed (Participants) | 1323 | 657
  Malaise (Post-injection 1) | 324 | 170
  Grade 3 Malaise (Post-injection 1): number analyzed (Participants) | 1323 | 657
  Grade 3 Malaise (Post-injection 1) | 32 | 15
  Myalgia (Post-injection 1): number analyzed (Participants) | 1323 | 657
  Myalgia (Post-injection 1) | 386 | 180
  Grade 3 Myalgia (Post-injection 1): number analyzed (Participants) | 1323 | 657
  Grade 3 Myalgia (Post-injection 1) | 29 | 10
  Asthenia (Post-injection 1): number analyzed (Participants) | 1323 | 657
  Asthenia (Post-injection 1) | 326 | 148
  Grade 3 Asthenia (Post-injection 1): number analyzed (Participants) | 1323 | 657
  Grade 3 Asthenia (Post-injection 1) | 36 | 17
  Fever (Post-injection 2): number analyzed (Participants) | 1228 | 594
  Fever (Post-injection 2) | 72 | 42
  Grade 3 Fever (Post-injection 2): number analyzed (Participants) | 1228 | 594
  Grade 3 Fever (Post-injection 2) | 10 | 7
  Headache (Post-injection 2): number analyzed (Participants) | 1297 | 639
  Headache (Post-injection 2) | 386 | 182
  Grade 3 Headache (Post-injection 2): number analyzed (Participants) | 1297 | 639
  Grade 3 Headache (Post-injection 2) | 27 | 15
  Malaise (Post-injection 2): number analyzed (Participants) | 1298 | 639
  Malaise (Post-injection 2) | 270 | 106
  Grade 3 Malaise (Post-injection 2): number analyzed (Participants) | 1298 | 639
  Grade 3 Malaise (Post-injection 2) | 17 | 8
  Myalgia (Post-injection 2): number analyzed (Participants) | 1298 | 639
  Myalgia (Post-injection 2) | 273 | 101
  Grade 3 Myalgia (Post-injection 2): number analyzed (Participants) | 1298 | 639
  Grade 3 Myalgia (Post-injection 2) | 21 | 5
  Asthenia (Post-injection 2): number analyzed (Participants) | 1298 | 639
  Asthenia (Post-injection 2) | 231 | 105
  Grade 3 Asthenia (Post-injection 2): number analyzed (Participants) | 1298 | 639
  Grade 3 Asthenia (Post-injection 2) | 24 | 7
  Fever (Post-injection 3): number analyzed (Participants) | 1215 | 597
  Fever (Post-injection 3) | 89 | 52
  Grade 3 Fever (Post-injection 3): number analyzed (Participants) | 1215 | 597
  Grade 3 Fever (Post-injection 3) | 13 | 5
  Headache (Post-injection 3): number analyzed (Participants) | 1277 | 631
  Headache (Post-injection 3) | 378 | 158
  Grade 3 Headache (Post-injection 3): number analyzed (Participants) | 1277 | 631
  Grade 3 Headache (Post-injection 3) | 33 | 12
  Malaise (Post-injection 3): number analyzed (Participants) | 1277 | 631
  Malaise (Post-injection 3) | 246 | 96
  Grade 3 Malaise (Post-injection 3): number analyzed (Participants) | 1277 | 631
  Grade 3 Malaise (Post-injection 3) | 18 | 7
  Myalgia (Post-injection 3): number analyzed (Participants) | 1277 | 631
  Myalgia (Post-injection 3) | 255 | 116
  Grade 3 Myalgia (Post-injection 3): number analyzed (Participants) | 1277 | 631
  Grade 3 Myalgia (Post-injection 3) | 19 | 5
  Asthenia (Post-injection 3): number analyzed (Participants) | 1277 | 631
  Asthenia (Post-injection 3) | 208 | 110
  Grade 3 Asthenia (Post-injection 3): number analyzed (Participants) | 1277 | 631
  Grade 3 Asthenia (Post-injection 3) | 17 | 8

ADVERSE EVENTS:
Time Frame: Unsolicited adverse event (AE) data were collected from Day 0 (post-vaccination) up to 28 days after each vaccination. Solicited Reaction (SR) data were collected within 7 and 14 days after vaccination. Serious adverse event (SAE) data were collected throughout the study (up to 72 months).
Description: Analysis were performed on Safety Analysis Set. A SR was an AE that was prelisted (i.e., solicited) in the electronic case report form (eCRF) and considered to be related to vaccination (adverse drug reaction). An unsolicited AE was an observed AE that did not fulfill the conditions prelisted (i.e., solicited) in the eCRF in terms of symptom and/or onset post-vaccination.
Groups:
- Placebo Group: Participants received 3 doses of placebo vaccine; one each at 0, 6, and 12 months.
Arm/Group | CYD Dengue Vaccine Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 42/13915 | 27/6939
Serious Adverse Events (participants affected / at risk) | 1765/13915 | 911/6939
Other Adverse Events (participants affected / at risk) | 1038/1333 | 515/664
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=13915) | Placebo Group (N=6939)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Anaemia Of Pregnancy (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Aplastic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Haemorrhagic Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 7 (7) | 4 (4)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymphoid Tissue Hyperplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Wolff-Parkinson-White Syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Arteriovenous Malformation (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Atrial Septal Defect (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Cryptorchism (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Hereditary Spherocytosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 3 (3)
Sickle Cell Trait (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Tympanic Membrane Perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Basedow's Disease (Endocrine disorders) | 1 (1) | 0 (0)
Hypothalamo-Pituitary Disorder (Endocrine disorders) | 1 (1) | 0 (0)
Keratoconus (Eye disorders) | 0 (0) | 1 (1)
Retinal Detachment (Eye disorders) | 1 (1) | 0 (0)
Visual Impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal Adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 26 (26) | 9 (9)
Abdominal Pain Lower (Gastrointestinal disorders) | 3 (3) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Acute Abdomen (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 4 (4)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (5) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 2 (3) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 2 (2) | 1 (1)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 12 (13) | 5 (5)
Gastritis Haemorrhagic (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 5 (5) | 2 (2)
Inguinal Hernia, Obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Functional Disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 1 (1)
Malocclusion (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 2 (2)
Peptic Ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Peritonitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical Hernia, Obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Varices Oesophageal (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting In Pregnancy (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter Site Phlebitis (General disorders) | 0 (0) | 1 (1)
Cyst (General disorders) | 0 (0) | 1 (1)
Death (General disorders) | 1 (1) | 0 (0)
Device Intolerance (General disorders) | 0 (0) | 1 (1)
Discomfort (General disorders) | 0 (0) | 1 (1)
Drowning (General disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 1 (1)
Medical Device Complication (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 9 (9) | 2 (2)
Soft Tissue Inflammation (General disorders) | 1 (1) | 0 (0)
Sudden Death (General disorders) | 2 (2) | 0 (0)
Autoimmune Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 7 (7) | 6 (6)
Cholecystitis Acute (Hepatobiliary disorders) | 5 (5) | 2 (2)
Cholecystitis Chronic (Hepatobiliary disorders) | 3 (3) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 9 (9) | 13 (15)
Cholestasis Of Pregnancy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Gallbladder Disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatitis Acute (Hepatobiliary disorders) | 2 (2) | 1 (1)
Hepatitis Toxic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hydrocholecystis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 2 (2)
Allergy To Arthropod Sting (Immune system disorders) | 1 (1) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Anti-Neutrophil Cytoplasmic Antibody Positive Vasculitis (Immune system disorders) | 1 (1) | 0 (0)
Antiphospholipid Syndrome (Immune system disorders) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 2 (2)
Food Allergy (Immune system disorders) | 0 (0) | 1 (1)
Abdominal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Abortion Infected (Infections and infestations) | 1 (1) | 2 (2)
Abscess (Infections and infestations) | 2 (2) | 0 (0)
Abscess Limb (Infections and infestations) | 6 (6) | 1 (1)
Abscess Neck (Infections and infestations) | 1 (1) | 1 (1)
Abscess Of Salivary Gland (Infections and infestations) | 0 (0) | 1 (1)
Abscess Oral (Infections and infestations) | 0 (0) | 2 (2)
Acute Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Acute Tonsillitis (Infections and infestations) | 1 (1) | 4 (4)
Adenoiditis (Infections and infestations) | 0 (0) | 1 (1)
Amniotic Cavity Infection (Infections and infestations) | 2 (3) | 1 (1)
Amoebiasis (Infections and infestations) | 0 (0) | 1 (1)
Amoebic Dysentery (Infections and infestations) | 2 (2) | 1 (1)
Anal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Anogenital Warts (Infections and infestations) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 261 (261) | 138 (138)
Appendicitis Perforated (Infections and infestations) | 5 (5) | 2 (2)
Arthritis Bacterial (Infections and infestations) | 3 (3) | 2 (2)
Arthritis Infective (Infections and infestations) | 1 (1) | 0 (0)
Asymptomatic Hiv Infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial Infection (Infections and infestations) | 3 (3) | 1 (1)
Bartholin's Abscess (Infections and infestations) | 2 (2) | 3 (3)
Breast Abscess (Infections and infestations) | 4 (4) | 3 (3)
Breast Cellulitis (Infections and infestations) | 6 (6) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 8 (8) | 0 (0)
Bronchopneumonia (Infections and infestations) | 6 (6) | 1 (1)
Carbuncle (Infections and infestations) | 1 (1) | 1 (1)
Cellulitis (Infections and infestations) | 50 (50) | 35 (35)
Chikungunya Virus Infection (Infections and infestations) | 8 (8) | 3 (3)
Chorioamnionitis (Infections and infestations) | 3 (3) | 2 (2)
Chronic Sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Chronic Tonsillitis (Infections and infestations) | 1 (1) | 2 (2)
Cutaneous Anthrax (Infections and infestations) | 2 (2) | 1 (1)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Dengue Fever (Infections and infestations) | 101 (104) | 94 (94)
Endometritis (Infections and infestations) | 3 (3) | 1 (1)
Endometritis Decidual (Infections and infestations) | 3 (3) | 2 (2)
Enterocolitis Infectious (Infections and infestations) | 1 (1) | 1 (1)
Erysipelas (Infections and infestations) | 2 (2) | 3 (3)
External Ear Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Eye Infection Toxoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Flavivirus Infection (Infections and infestations) | 3 (3) | 0 (0)
Gastroenteritis (Infections and infestations) | 34 (34) | 21 (21)
Gastroenteritis Bacterial (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 3 (3) | 2 (2)
Gastrointestinal Bacterial Infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal Infection (Infections and infestations) | 3 (3) | 1 (1)
Gastrointestinal Viral Infection (Infections and infestations) | 0 (0) | 1 (1)
Genital Infection Female (Infections and infestations) | 1 (1) | 0 (0)
Genitourinary Tract Infection (Infections and infestations) | 0 (0) | 2 (2)
Granuloma Inguinale (Infections and infestations) | 1 (1) | 0 (0)
H1n1 Influenza (Infections and infestations) | 1 (1) | 0 (0)
Hiv Infection (Infections and infestations) | 2 (2) | 1 (1)
Hiv Infection Cdc Category A3 (Infections and infestations) | 1 (1) | 0 (0)
Helminthic Infection (Infections and infestations) | 1 (1) | 1 (1)
Hepatitis A (Infections and infestations) | 3 (3) | 1 (1)
Hepatitis Viral (Infections and infestations) | 2 (2) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 1 (1)
Herpes Zoster Ophthalmic (Infections and infestations) | 0 (0) | 1 (1)
Infected Bites (Infections and infestations) | 1 (1) | 1 (1)
Infectious Mononucleosis (Infections and infestations) | 2 (2) | 1 (1)
Infective Myositis (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 1 (1)
Leptospirosis (Infections and infestations) | 2 (2) | 1 (1)
Lower Respiratory Tract Infection (Infections and infestations) | 2 (2) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 0 (0) | 1 (1)
Mastitis (Infections and infestations) | 4 (4) | 3 (3)
Mastitis Postpartum (Infections and infestations) | 1 (1) | 3 (3)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis Bacterial (Infections and infestations) | 2 (2) | 1 (1)
Meningitis Viral (Infections and infestations) | 1 (1) | 1 (1)
Mononucleosis Syndrome (Infections and infestations) | 1 (1) | 0 (0)
Mumps (Infections and infestations) | 0 (0) | 1 (1)
Mycoplasma Infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Orchitis (Infections and infestations) | 5 (5) | 2 (2)
Osteomyelitis (Infections and infestations) | 2 (3) | 1 (1)
Osteomyelitis Chronic (Infections and infestations) | 4 (4) | 1 (1)
Otitis Media (Infections and infestations) | 0 (0) | 2 (2)
Otitis Media Chronic (Infections and infestations) | 0 (0) | 1 (2)
Pancreatitis Mumps (Infections and infestations) | 1 (1) | 0 (0)
Panencephalitis (Infections and infestations) | 0 (0) | 1 (1)
Parasitic Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Pelvic Inflammatory Disease (Infections and infestations) | 10 (11) | 4 (4)
Perineal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Perineal Infection (Infections and infestations) | 0 (0) | 1 (1)
Periorbital Cellulitis (Infections and infestations) | 2 (2) | 1 (1)
Peritonsillar Abscess (Infections and infestations) | 2 (2) | 2 (2)
Pharyngotonsillitis (Infections and infestations) | 3 (3) | 0 (0)
Pilonidal Cyst (Infections and infestations) | 5 (6) | 1 (1)
Pneumonia (Infections and infestations) | 18 (18) | 13 (13)
Pneumonia Bacterial (Infections and infestations) | 4 (4) | 0 (0)
Pneumonia Mycoplasmal (Infections and infestations) | 1 (1) | 0 (0)
Post Procedural Infection (Infections and infestations) | 1 (1) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 6 (8) | 4 (4)
Postpartum Sepsis (Infections and infestations) | 4 (4) | 0 (0)
Pulmonary Tuberculosis (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis (Infections and infestations) | 10 (12) | 0 (0)
Pyelonephritis Acute (Infections and infestations) | 7 (7) | 1 (1)
Retroperitoneal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Salmonellosis (Infections and infestations) | 2 (2) | 0 (0)
Scarlet Fever (Infections and infestations) | 0 (0) | 1 (1)
Secondary Syphilis (Infections and infestations) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Skin Infection (Infections and infestations) | 1 (1) | 0 (0)
Soft Tissue Infection (Infections and infestations) | 1 (1) | 0 (0)
Subcutaneous Abscess (Infections and infestations) | 13 (13) | 2 (2)
Syphilis (Infections and infestations) | 2 (2) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 2 (2)
Tonsillitis Bacterial (Infections and infestations) | 2 (2) | 1 (1)
Tooth Abscess (Infections and infestations) | 6 (6) | 2 (3)
Toxoplasmosis (Infections and infestations) | 0 (0) | 2 (2)
Tracheitis (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Typhoid Fever (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 118 (127) | 59 (69)
Urinary Tract Infection Bacterial (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Vaginal Infection (Infections and infestations) | 1 (1) | 1 (1)
Varicella (Infections and infestations) | 3 (3) | 1 (1)
Viral Cardiomyopathy (Infections and infestations) | 1 (1) | 0 (0)
Viral Infection (Infections and infestations) | 10 (10) | 7 (7)
Visceral Leishmaniasis (Infections and infestations) | 1 (1) | 0 (0)
Vulval Abscess (Infections and infestations) | 1 (1) | 1 (1)
Wound Infection (Infections and infestations) | 5 (5) | 0 (0)
Abdominal Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Accident At Home (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Accident At Work (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Acetabulum Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Adverse Event Following Immunisation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Animal Bite (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Ankle Fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Arthropod Sting (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Avulsion Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Burns Second Degree (Injury, poisoning and procedural complications) | 6 (6) | 2 (2)
Burns Third Degree (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Chemical Poisoning (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Chest Injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Endotracheal Intubation Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Epiphyseal Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye Injury (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Eye Penetration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 28 (28) | 11 (12)
Femur Fracture (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Fibula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Forearm Fracture (Injury, poisoning and procedural complications) | 21 (21) | 7 (7)
Foreign Body (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Foreign Body In Eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Genital Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gun Shot Wound (Injury, poisoning and procedural complications) | 24 (24) | 15 (15)
Hand Fracture (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Head Injury (Injury, poisoning and procedural complications) | 16 (17) | 3 (3)
Humerus Fracture (Injury, poisoning and procedural complications) | 6 (6) | 5 (5)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional Overdose (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Joint Injury (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Limb Crushing Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Limb Traumatic Amputation (Injury, poisoning and procedural complications) | 4 (4) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 3 (3) | 3 (3)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus Lesion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Multiple Fractures (Injury, poisoning and procedural complications) | 6 (6) | 1 (1)
Multiple Injuries (Injury, poisoning and procedural complications) | 12 (12) | 3 (3)
Muscle Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Nerve Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Open Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Perineal Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Poisoning Deliberate (Injury, poisoning and procedural complications) | 15 (16) | 10 (10)
Post Procedural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post-Traumatic Pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative Wound Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius Fracture (Injury, poisoning and procedural complications) | 8 (8) | 3 (3)
Road Traffic Accident (Injury, poisoning and procedural complications) | 108 (109) | 39 (39)
Skull Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft Tissue Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal Cord Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal Cord Injury Cervical (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Sports Injury (Injury, poisoning and procedural complications) | 8 (8) | 3 (3)
Stab Wound (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Tendon Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon Rupture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Testicular Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia Fracture (Injury, poisoning and procedural complications) | 5 (5) | 3 (3)
Toxicity To Various Agents (Injury, poisoning and procedural complications) | 7 (7) | 4 (4)
Traumatic Brain Injury (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ulna Fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Ulnar Nerve Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vascular Access Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 5 (5) | 2 (2)
Wrist Fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Investigation (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 1 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Ankle Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthropathy (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Epiphysiolysis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Juvenile Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Knee Deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rheumatic Fever (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Systemic Lupus Erythematosus (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Benign Hydatidiform Mole (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Benign Ovarian Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign Pancreatic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone Giant Cell Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bone Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Chronic Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Desmoid Tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Fibroadenoma Of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Haemangioma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Osteoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Osteosarcoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Osteosarcoma Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Ovarian Germ Cell Teratoma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Acute Disseminated Encephalomyelitis (Nervous system disorders) | 0 (0) | 1 (1)
Acute Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Arachnoid Cyst (Nervous system disorders) | 1 (1) | 0 (0)
Atonic Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Cerebellar Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Complicated Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Convulsion (Nervous system disorders) | 21 (31) | 10 (11)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Encephalitis (Nervous system disorders) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 26 (86) | 8 (27)
Grand Mal Convulsion (Nervous system disorders) | 2 (2) | 2 (4)
Guillain-Barre Syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1) | 1 (1)
Haemorrhagic Cerebral Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Hydrocephalus (Nervous system disorders) | 1 (1) | 0 (0)
Hypersomnia (Nervous system disorders) | 0 (0) | 1 (1)
Hypertensive Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Idiopathic Generalised Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Intracranial Aneurysm (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 5 (5) | 2 (2)
Migraine With Aura (Nervous system disorders) | 0 (0) | 1 (1)
Migraine Without Aura (Nervous system disorders) | 2 (2) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 0 (0) | 1 (1)
Partial Seizures (Nervous system disorders) | 1 (1) | 1 (1)
Post-Traumatic Headache (Nervous system disorders) | 1 (1) | 0 (0)
Status Epilepticus (Nervous system disorders) | 3 (3) | 1 (3)
Status Migrainosus (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 6 (6) | 2 (2)
Viith Nerve Paralysis (Nervous system disorders) | 5 (5) | 3 (3)
Abnormal Product Of Conception (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion (Pregnancy, puerperium and perinatal conditions) | 14 (14) | 6 (6)
Abortion Complete (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 4 (4)
Abortion Complicated (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion Incomplete (Pregnancy, puerperium and perinatal conditions) | 22 (22) | 9 (9)
Abortion Incomplete Complicated (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion Missed (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2)
Abortion Of Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 48 (51) | 30 (34)
Abortion Spontaneous Complete (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 6 (6)
Abortion Spontaneous Complicated (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Abortion Spontaneous Incomplete (Pregnancy, puerperium and perinatal conditions) | 16 (16) | 2 (2)
Abortion Spontaneous Incomplete Complicated (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion Threatened (Pregnancy, puerperium and perinatal conditions) | 14 (14) | 3 (4)
Amniorrhexis (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Antepartum Haemorrhage (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Blighted Ovum (Pregnancy, puerperium and perinatal conditions) | 11 (11) | 1 (1)
Cephalo-Pelvic Disproportion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Cervical Incompetence (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Complication Of Delivery (Pregnancy, puerperium and perinatal conditions) | 4 (4) | 0 (0)
Delivery (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 0 (0)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3)
Failed Induction Of Labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
False Labour (Pregnancy, puerperium and perinatal conditions) | 39 (45) | 14 (14)
Foetal Distress Syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 4 (4)
Gestational Hypertension (Pregnancy, puerperium and perinatal conditions) | 12 (12) | 7 (7)
Hellp Syndrome (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
High Risk Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Hyperemesis Gravidarum (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0)
Intra-Uterine Death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3)
Intrapartum Haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 12 (12) | 4 (4)
Placental Insufficiency (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Postpartum Haemorrhage (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 5 (5)
Pre-Eclampsia (Pregnancy, puerperium and perinatal conditions) | 34 (35) | 23 (23)
Premature Baby (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Premature Delivery (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 1 (1)
Premature Labour (Pregnancy, puerperium and perinatal conditions) | 17 (17) | 6 (6)
Premature Rupture Of Membranes (Pregnancy, puerperium and perinatal conditions) | 13 (13) | 2 (2)
Premature Separation Of Placenta (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Prolonged Labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3)
Puerperal Pyrexia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Retained Placenta Or Membranes (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2)
Retained Products Of Conception (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1)
Ruptured Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 6 (6) | 5 (5)
Threatened Labour (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 9 (10)
Abnormal Behaviour (Psychiatric disorders) | 1 (1) | 0 (0)
Acute Psychosis (Psychiatric disorders) | 2 (2) | 1 (1)
Acute Stress Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Adjustment Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 1 (1)
Anorexia Nervosa (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety Disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Bipolar I Disorder (Psychiatric disorders) | 2 (4) | 0 (0)
Bipolar Disorder (Psychiatric disorders) | 2 (2) | 3 (3)
Completed Suicide (Psychiatric disorders) | 2 (2) | 2 (2)
Conduct Disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Conversion Disorder (Psychiatric disorders) | 3 (3) | 1 (1)
Dependence (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 18 (18) | 9 (9)
Depression Suicidal (Psychiatric disorders) | 0 (0) | 2 (2)
Dissociative Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Drug Abuse (Psychiatric disorders) | 2 (2) | 1 (1)
Drug Dependence (Psychiatric disorders) | 1 (1) | 0 (0)
Intentional Drug Misuse (Psychiatric disorders) | 1 (1) | 1 (1)
Intentional Self-Injury (Psychiatric disorders) | 6 (6) | 2 (2)
Intermittent Explosive Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 6 (6) | 2 (2)
Obsessive Rumination (Psychiatric disorders) | 0 (0) | 1 (1)
Psychotic Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 1 (1) | 2 (2)
Schizophrenia, Undifferentiated Type (Psychiatric disorders) | 1 (1) | 0 (0)
Somatoform Disorder (Psychiatric disorders) | 1 (1) | 1 (1)
Substance Abuse (Psychiatric disorders) | 14 (15) | 9 (13)
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 19 (19) | 8 (14)
Calculus Ureteric (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus Urethral (Renal and urinary disorders) | 1 (1) | 0 (0)
Calculus Urinary (Renal and urinary disorders) | 3 (3) | 1 (1)
Cystitis Haemorrhagic (Renal and urinary disorders) | 0 (0) | 1 (1)
Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Lupus Nephritis (Renal and urinary disorders) | 1 (1) | 1 (1)
Nephritic Syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 15 (15) | 5 (5)
Post Streptococcal Glomerulonephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Colic (Renal and urinary disorders) | 2 (2) | 3 (5)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Tubular Necrosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Tubulointerstitial Nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urogenital Haemorrhage (Renal and urinary disorders) | 1 (1) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Balanitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Bartholinitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast Disorder (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Breast Mass (Reproductive system and breast disorders) | 4 (4) | 1 (1)
Breast Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Coital Bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 3 (5) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Endometriosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Female Genital Tract Fistula (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Haematocolpos (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Haematosalpinx (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Haemorrhagic Ovarian Cyst (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian Cyst (Reproductive system and breast disorders) | 7 (7) | 5 (5)
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Ovarian Torsion (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovulation Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Polycystic Ovaries (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Retrograde Menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular Disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Testicular Torsion (Reproductive system and breast disorders) | 12 (12) | 3 (3)
Uterine Cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine Haemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal Haemorrhage (Reproductive system and breast disorders) | 3 (3) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vulval Haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Adenoidal Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Alveolitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 19 (24) | 17 (22)
Asthmatic Crisis (Respiratory, thoracic and mediastinal disorders) | 12 (14) | 7 (8)
Bronchial Obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal Turbinate Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary Artery Stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Tract Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Status Asthmaticus (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 2 (2)
Tonsillar Cyst (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis Atopic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Henoch-Schonlein Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertrophic Scar (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Mechanical Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin Fissures (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Subcutaneous Nodule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Physical Assault (Social circumstances) | 9 (9) | 4 (4)
Sexual Abuse (Social circumstances) | 7 (7) | 4 (4)
Substance Use (Social circumstances) | 1 (1) | 0 (0)
Victim Of Crime (Social circumstances) | 2 (2) | 0 (0)
Victim Of Homicide (Social circumstances) | 5 (5) | 1 (1)
Victim Of Sexual Abuse (Social circumstances) | 1 (1) | 1 (1)
Abortion Induced (Surgical and medical procedures) | 0 (0) | 1 (1)
Abortion Induced Complete (Surgical and medical procedures) | 1 (1) | 0 (0)
Caesarean Section (Surgical and medical procedures) | 2 (2) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Obesity Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Scoliosis Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Umbilical Hernia Repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 0 (0)
Secondary Hypertension (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=1333) | Placebo Group (N=664)
Asthenia (General disorders) | 500 (771) | 253 (366)
Injection Site Erythema (General disorders) | 83 (99) | 44 (52)
Injection Site Pain (General disorders) | 650 (1056) | 270 (384)
Injection Site Swelling (General disorders) | 77 (92) | 27 (32)
Malaise (General disorders) | 539 (853) | 264 (383)
Pyrexia (General disorders) | 238 (270) | 127 (142)
Influenza (Infections and infestations) | 76 (80) | 37 (40)
Nasopharyngitis (Infections and infestations) | 150 (163) | 60 (70)
Myalgia (Musculoskeletal and connective tissue disorders) | 578 (921) | 267 (400)
Headache (Nervous system disorders) | 753 (1385) | 388 (652)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.